CLINICAL TRIAL: NCT04952376
Title: Enabling Equitable Access to COVID-19 Vaccine in Under-Resourced Communities
Brief Title: Equitable Access to COVID-19 Vaccines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Adelante Healthcare (Unknown)
Responsible Party: Principal Investigator, Chyke A. Doubeni, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-002939
Record Dates: First submitted 2021-06-07; First posted 2021-07-07 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Drug Interactions

STUDY DESIGN:
Intervention Model Description: Arm 1: Patient is informed via SMS of vaccine availability and advised to schedule an appointment.
  Arm 2: Same as Arm 1 but delivered as a personalized message text from the PCP. Arm 3: Patients assigned to Arm 3 will receive the same message in the Arm 2 intervention. In addition, they will be given interactive or 2-way SMS options to obtain additional information about COVID vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short message service (SMS) (Active Comparator): Subjects will receive vaccine availability and appointment information via SMS.
  Interventions: Behavioral: SMS delivery of information
- Personalized text message (Experimental): Subjects will receive vaccine availability and appointment information via a personalized message text from the primary care provider (PCP).
  Interventions: Behavioral: Personalized text message delivery of information
- Interactive or 2-way SMS (Experimental): Subjects will receive vaccine availability and appointment information via interactive 2-way SMS options.
  Interventions: Behavioral: Interactive or 2-way SMS delivery of information

INTERVENTIONS:
Behavioral: SMS delivery of information — Patients are informed via SMS that COVID-19 vaccine doses are available and advised to schedule an appointment. Links to information or phone for scheduling will be provided. Messages mimic the clinic's usual practice of information delivery to patients
  Arms: Short message service (SMS)
Behavioral: Personalized text message delivery of information — Patients are informed via SMS that COVID-19 vaccine doses are available and advised to schedule an appointment. The SMS message is personalized as a recommendation from the primary care clinician
  Arms: Personalized text message
Behavioral: Interactive or 2-way SMS delivery of information — This intervention is same as in the Arm 2 using personalized messaging from the PCP. In addition, patients are given interactive or 2-way SMS options to obtain additional information about COVID vaccine and answers to frequently asked questions.
  Arms: Interactive or 2-way SMS

SUMMARY:
This study will deploy a multimodal pragmatic intervention to improve vaccine uptake in priority populations and address vaccine hesitancy to improve access by using a proactive organized population-based outreach leveraging health information technology with tailored navigation support to address mistrust and social barriers.

DETAILED DESCRIPTION:
This study will deploy a multimodal pragmatic intervention to improve vaccine uptake in priority populations through a proactive organized population-based outreach approach. It will leverage health information technology with tailored navigation support to address mistrust and social barriers. Study key objectives are to:

1. conduct a survey of patients to assess and track barriers, intent, and sources of information on COVID vaccine over time.
2. Determine whether a primary care physician (PCP) endorsement with or without interactive digital communication plus navigation is more effective in promoting uptake of COVID-19 vaccine than general messages from the clinic. Patients will be randomized to one of three arms:

   1. Arm 1: Message about vaccine availability delivered by SMS advising patients to make an appointment.
   2. Arm 2: Same as Arm 1 but delivered as a personalized message text from the PCP.
   3. Arm 3: Same as Arm 2 plus a interactive 2-way SMS options.

ELIGIBILITY:
Inclusion Criteria: 18 years and older, receiving care at Adelante Healthcare and not vaccinated or already scheduled for vaccination through the health center's appointment system Exclusion Criteria: Patient younger than 18 or who have been previously or are selected for vaccination during or prior to the week of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1722 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Dose 1 COVID-19 Vaccine | 30 days
  Primary outcome will be the receipt of the first dose of any of the COVID-19 vaccines with FDA emergency use authorization

SECONDARY OUTCOMES:
Dose 2 COVID-19 Vaccine | 60 days
  Examine receipt of all doses as recommended by the manufacturer (for most vaccine2 doses).

OTHER OUTCOMES:
Engagement | 30 days
  We will assess engagement with the 2-way SMS options as well as use of online appointment scheduling

CONTACTS AND LOCATIONS:
Overall Officials: Chyke Doubeni, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials